CLINICAL TRIAL: NCT00192374
Title: A Prospective, Randomized, Double-Blind, Placebo-Controlled, Phase III, Multicenter Trial to Compare the Safety, Tolerability, Immunogenicity and Efficacy of Three Dose Levels of a Liquid Formulation of Influenza Virus Vaccine, Trivalent, Types A & B,Live, Cold-Adapted (CAIV-T) in Healthy Children
Brief Title: Trial to Compare the Safety, Tolerability, Immunogenicity and Efficacy of Three Dose Levels of a Liquid Formulation of Influenza Virus Vaccine, (CAIV-T) in Healthy Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: D153-P513
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2006-10-03 (Estimated); Status verified 2006-10

CONDITIONS: Healthy
MeSH Terms: interventions — Fluid Therapy

INTERVENTIONS:
Biological: CAIV-T, Liquid

SUMMARY:
- Trial to Compare the Safety, Tolerability, Immunogenicity and Efficacy of Three Dose Levels of a Liquid Formulation of(CAIV-T) in Healthy Children.

DETAILED DESCRIPTION:
- A Prospective, Randomized, Double-Blind, Placebo-Controlled, Phase III, Multicenter Trial to Compare the Safety, Tolerability, Immunogenicity and Efficacy of Three Dose Levels of a Liquid Formulation of Influenza Virus Vaccine, Trivalent, Types A & B, Live Cold-Adapted (CAIV-T) in Healthy Children

ELIGIBILITY:
Inclusion Criteria:

* •who are aged at least 6 months and less than 36 months of age at the time of first vaccination

  * who are in good health as determined by medical history, physical examination and clinical judgement
  * whose parent(s)/legal guardian(s) have provided written informed consent after the nature of the study has been explained
  * who, along with their parent(s)/legal guardian(s), will be available for duration of the trial (8 months ±1 month)
  * whose parent(s)/legal guardian(s), can be reached by study staff for the post-vaccination contacts [telephone, clinic or home visit].

Exclusion Criteria:

* whose parent(s)/legal guardian(s) are perceived to be unavailable or difficult to contact for evaluation or study visits during the study period with any serious chronic disease (e.g., with signs of cardiac or renal failure or severe malnutrition), including progressive neurological disease

  * with Down's syndrome or other known cytogenetic disorders
  * with a known or suspected disease of the immune system or those receiving immunosuppressive therapy, including systemic corticosteroids (see Section 4.2.1)
  * who received any blood products, including immunoglobulin, in the period from six months prior to vaccination through to the conclusion of the study
  * for whom there is intent to administer any other investigational vaccine or agent from one month prior to enrollment through to the conclusion of the study
  * have an immunosuppressed or an immunocompromised individual living in the same household
  * who, at any time prior to entry into this study, received a dose of any influenza vaccine (commercial or investigational)
  * with a documented history of hypersensitivity to egg or egg protein or any other component of the assigned study vaccine
  * who received aspirin (acetylsalicylic acid) or aspirin-containing products in the two weeks prior to vaccination or for which use is anticipated during the study
  * with any medical conditions that in the opinion of the investigator might interfere with interpretation of the study results. If any of these criteria are met following enrolment, the subject will be excluded from subsequent vaccine dosing.

Note: Pregnancy in a household member or any person who has regular contact with the subject is not a contraindication to the enrollment or ongoing participation of the subject in the study.

Ages: 6 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1920
Dates: Start 2002-02; Study Completion 2002-11

PRIMARY OUTCOMES:
The primary efficacy endpoint was the first episode in a study child of a culture-confirmed influenza illness, caused by community-acquired subtypes antigenically similar to those contained in the vaccine.

SECONDARY OUTCOMES:
A secondary efficacy endpoint was the first episode of culture-confirmed influenza illness caused by any community-acquired antigenic subtype.

CONTACTS AND LOCATIONS:
Overall Officials: Tawee Chotpitayasunondh, Dr., Principal Investigator — Queen Sirikit National Institute of Child Health (Children's Hospital); Rosario Z. Capeding, Dr., Principal Investigator — Department of Microbiology, Research Institute for Tropical Medicine
Locations (2):
- Department of Microbiology, Research Institute for Tropical Medicine, City of Muntinlupa, Philippines
- Queen Sirikit National Institute of Child Health (Children's Hospital), Bangkok, Thailand